CLINICAL TRIAL: NCT00899782
Title: The CALGB Lung Cancer Tissue Bank
Brief Title: Collection and Storage of Blood and Tissue Samples From Patients Who Are Undergoing Surgery For Lung Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-140202; CALGB-140202; CDR0000271323 (Registry Identifier: NCI Physician Data Query); U10CA031946 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Lung Carcinoma; Lung Neoplasm; Malignant Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (lung cancer tissue bank): Grossly viable tumor and grossly normal lung tissue are identified and removed from patient surgical specimens and cryopreserved until shipment to the CALGB Lung Cancer Tissue Bank for future use in research. Blood specimens are also collected prior to surgery and at 4-12 weeks post-surgery (before the start of adjuvant therapy) and shipped immediately to the Tissue Bank.
  Interventions: Other: cytology specimen collection procedure

INTERVENTIONS:
Other: cytology specimen collection procedure — correlative studies
  Other Names: cytologic sampling

SUMMARY:
This research studies collecting and storing tissue and blood samples from patients with lung cancer who are undergoing surgery. Collecting and storing samples of tissue and blood from patients with lung cancer to study in the laboratory may help doctors learn more about changes that may occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To collect, catalog and store frozen samples of lung carcinoma and when possible, portions of involved lymph nodes, as well as adjacent grossly uninvolved lung tissue obtained from surgical specimens of patients undergoing surgical resection for previously untreated lung cancer as a source of quality DNA, messenger ribonucleic acid (mRNA) and protein for molecular analysis.
2. To collect, catalog and store frozen samples of blood pre- and post-resection from the same patients to provide a source of reference DNA to assess somatic mutations associated with tumor or preneoplastic "normal" lung, and to allow assessment of levels of circulating markers.
3. To associate these specimens with historical, clinical, pathological, and outcome information.

Grossly viable tumor and grossly normal lung tissue are identified and removed from patient surgical specimens and cryopreserved until shipment to the Cancer and Leukemia Group B (CALGB) Lung Cancer Tissue Bank for future use in research. Blood specimens are also collected prior to surgery and at 4-12 weeks post-surgery (before the start of adjuvant therapy) and shipped immediately to the Tissue Bank.

ELIGIBILITY:
1. Histologic Documentation: All patients with suspected or histologically documented previously untreated lung cancer undergoing surgical resection are eligible whether or not the patient participates in a CALGB-sponsored treatment trial; patients enrolled on a CALGB trial of preoperative chemotherapy for lung cancer will be eligible if a pre-treatment frozen sample of tumor (e.g., a positive lymph node from mediastinoscopy) can be submitted to the bank; patients enrolled on CALGB 140203, intraoperative sentinel node mapping in non-small cell lung cancer, are not eligible.
2. No patients with known infectious disease, such as human immunodeficiency virus (HIV), tuberculosis (TB), or hepatitis B, C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or histologically documented previously untreated lung cancer undergoing surgical resection at a CALGB Lung Cancer Tissue Bank-approved institution.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-07-15 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Collection and storage of frozen tissue samples for molecular analysisor resection of lung cancer | Up to 5 years
Collection and storage of frozen blood samples for the assessment of somatic mutations and levels of circulating markersto assess levels of circulating markers | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William Richards, MD, Study Chair — Brigham and Women's Cancer Center
Locations (19):
- United States (19):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Union Hospital of Cecil County, Elkton, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont